CLINICAL TRIAL: NCT01344759
Title: Effect of Increasing Depth of Dexmedetomidine and Propofol Anesthesia on Upper Airway Morphology in Children With History of Obstructive Sleep Apnea
Brief Title: Dexmedetomidine and Propofol in Children With History of Obstructive Sleep Apnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCHMC 2009-0514
Record Dates: First submitted 2011-04-21; First posted 2011-04-29 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea; MRI; Pediatrics; Dexmedetomidine; Propofol; Anesthesia
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator)
  Interventions: Drug: Propofol
- Dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Once an IV is in place, atropine 10 mcg/kg will be given. Loading dose of dexmedetomidine 1 mcg/kg will be administered over 10 minutes followed by a continuous infusion of dexmedetomidine at rate of 1 mcg/kg/h using a syringe pump.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Propofol — Once an IV is in place, atropine 10 mcg/kg will be given. Loading dose of propofol 2 mg/kg will be administered over 2 minutes followed by a continuous infusion of propofol at rate of 100 mcg/kg/minute using a syringe pump.
  Other Names: Diprivan
  Arms: Propofol

SUMMARY:
The purpose of this research study is to examine the effects of two commonly used anesthetic drugs, dexmedetomidine and propofol, have on the shape and muscle tone of the upper airway in children, adolescents, and young adults with a history of obstructive sleep apnea (OSA) having an MRI scan.

The results of this study will help in making the best decisions regarding the anesthesia medications that are most appropriate for children, adolescents, and young adults with OSA during MRI studies.

DETAILED DESCRIPTION:
Patients with OSA are at risk for airway obstruction (a condition that makes it difficult to breath) during sedation and anesthesia. Dexmedetomidine and propofol are safe and effective drugs regularly used by anesthesiologists. These drugs are used to put patients to sleep for operations and certain studies like MRI scans. However, there have been no studies describing the effects these drugs have on the upper airway of children, adolescents, and young adults with OSA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented history of OSA by polysomnography who require anesthesia for MRI sleep study or MRI brain imaging study.
2. Subjects must be 12 months to 25 years of age (inclusive)
3. Either the subject (if subject's age is 18-25) or the subject's legally authorized representative has given written informed consent to participate in the study

Exclusion Criteria:

1. The subject has life-threatening medical conditions (American Society of Anesthesiologists Physical Status 4, 5 or 6). The American Society of Anesthesiologists (ASA) classification scale is a measure of physical status or how healthy the patient is. For our study, we will focus on children which are defined as ASA I, II or III which means a healthy child (ASA I), a child with a systemic disease that is mild and well controlled (ASA II) or a child with systemic disease that is severe and controlled (ASA III).
2. The subject is allergic to or has a contraindication to propofol or dexmedetomidine.
3. The subject has a tracheostomy or other mechanical airway device
4. The subject is not scheduled to receive anesthesia-sedation care for the MRI
5. The subject has a history or a family (parent or sibling) history of malignant hyperthermia.

Ages: 12 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mahmoud, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Mason KP, Zgleszewski SE, Dearden JL, Dumont RS, Pirich MA, Stark CD, D'Angelo P, Macpherson S, Fontaine PJ, Connor L, Zurakowski D. Dexmedetomidine for pediatric sedation for computed tomography imaging studies. Anesth Analg. 2006 Jul;103(1):57-62, table of contents. doi: 10.1213/01.ane.0000216293.16613.15. PMID 16790626
- [Background] Ebert TJ, Hall JE, Barney JA, Uhrich TD, Colinco MD. The effects of increasing plasma concentrations of dexmedetomidine in humans. Anesthesiology. 2000 Aug;93(2):382-94. doi: 10.1097/00000542-200008000-00016. PMID 10910487
- [Background] Talke P, Lobo E, Brown R. Systemically administered alpha2-agonist-induced peripheral vasoconstriction in humans. Anesthesiology. 2003 Jul;99(1):65-70. doi: 10.1097/00000542-200307000-00014. PMID 12826844
- [Background] Talke P, Richardson CA, Scheinin M, Fisher DM. Postoperative pharmacokinetics and sympatholytic effects of dexmedetomidine. Anesth Analg. 1997 Nov;85(5):1136-42. doi: 10.1097/00000539-199711000-00033. PMID 9356115
- [Background] Doze VA, Chen BX, Maze M. Dexmedetomidine produces a hypnotic-anesthetic action in rats via activation of central alpha-2 adrenoceptors. Anesthesiology. 1989 Jul;71(1):75-9. doi: 10.1097/00000542-198907000-00014. PMID 2568769
- [Background] Drummond GB. Comparison of sedation with midazolam and ketamine: effects on airway muscle activity. Br J Anaesth. 1996 May;76(5):663-7. doi: 10.1093/bja/76.5.663. PMID 8688266
- [Background] Drummond GB. Influence of thiopentone on upper airway muscles. Br J Anaesth. 1989 Jul;63(1):12-21. doi: 10.1093/bja/63.1.12. PMID 2765337
- [Background] Hwang JC, St John WM, Bartlett D Jr. Respiratory-related hypoglossal nerve activity: influence of anesthetics. J Appl Physiol Respir Environ Exerc Physiol. 1983 Sep;55(3):785-92. doi: 10.1152/jappl.1983.55.3.785. PMID 6629915
- [Background] Hudgel DW, Harasick T, Katz RL, Witt WJ, Abelson TI. Uvulopalatopharyngoplasty in obstructive apnea. Value of preoperative localization of site of upper airway narrowing during sleep. Am Rev Respir Dis. 1991 May;143(5 Pt 1):942-6. doi: 10.1164/ajrccm/143.5_Pt_1.942. PMID 2024847
- [Background] Nandi PR, Charlesworth CH, Taylor SJ, Nunn JF, Dore CJ. Effect of general anaesthesia on the pharynx. Br J Anaesth. 1991 Feb;66(2):157-62. doi: 10.1093/bja/66.2.157. PMID 1817614
- [Background] SAFAR P, ESCARRAGA LA, CHANG F. Upper airway obstruction in the unconscious patient. J Appl Physiol. 1959 Sep;14:760-4. doi: 10.1152/jappl.1959.14.5.760. No abstract available. PMID 14440737
- [Background] Litman RS, Kottra JA, Berkowitz RJ, Ward DS. Upper airway obstruction during midazolam/nitrous oxide sedation in children with enlarged tonsils. Pediatr Dent. 1998 Sep-Oct;20(5):318-20. PMID 9803430
- [Background] Donnelly LF, Casper KA, Chen B, Koch BL. Defining normal upper airway motion in asymptomatic children during sleep by means of cine MR techniques. Radiology. 2002 Apr;223(1):176-80. doi: 10.1148/radiol.2231011023. PMID 11930064
- [Background] Donnelly LF, Shott SR, LaRose CR, Chini BA, Amin RS. Causes of persistent obstructive sleep apnea despite previous tonsillectomy and adenoidectomy in children with down syndrome as depicted on static and dynamic cine MRI. AJR Am J Roentgenol. 2004 Jul;183(1):175-81. doi: 10.2214/ajr.183.1.1830175. PMID 15208134
- [Background] Ibacache ME, Munoz HR, Brandes V, Morales AL. Single-dose dexmedetomidine reduces agitation after sevoflurane anesthesia in children. Anesth Analg. 2004 Jan;98(1):60-63. doi: 10.1213/01.ANE.0000094947.20838.8E. PMID 14693585
- [Background] Guler G, Akin A, Tosun Z, Ors S, Esmaoglu A, Boyaci A. Single-dose dexmedetomidine reduces agitation and provides smooth extubation after pediatric adenotonsillectomy. Paediatr Anaesth. 2005 Sep;15(9):762-6. doi: 10.1111/j.1460-9592.2004.01541.x. PMID 16101707
- [Background] Petroz GC, Sikich N, James M, van Dyk H, Shafer SL, Schily M, Lerman J. A phase I, two-center study of the pharmacokinetics and pharmacodynamics of dexmedetomidine in children. Anesthesiology. 2006 Dec;105(6):1098-110. doi: 10.1097/00000542-200612000-00009. PMID 17122572
- [Background] Mahmoud M, Tyler T, Sadhasivam S. Dexmedetomidine and ketamine for large anterior mediastinal mass biopsy. Paediatr Anaesth. 2008 Oct;18(10):1011-3. doi: 10.1111/j.1460-9592.2008.02604.x. No abstract available. PMID 18811855
- [Background] Eastwood PR, Platt PR, Shepherd K, Maddison K, Hillman DR. Collapsibility of the upper airway at different concentrations of propofol anesthesia. Anesthesiology. 2005 Sep;103(3):470-7. doi: 10.1097/00000542-200509000-00007. PMID 16129969
- [Background] Mason KP, Zurakowski D, Zgleszewski SE, Robson CD, Carrier M, Hickey PR, Dinardo JA. High dose dexmedetomidine as the sole sedative for pediatric MRI. Paediatr Anaesth. 2008 May;18(5):403-11. doi: 10.1111/j.1460-9592.2008.02468.x. Epub 2008 Mar 18. PMID 18363626
- [Background] Mason KP, Zgleszewski SE, Prescilla R, Fontaine PJ, Zurakowski D. Hemodynamic effects of dexmedetomidine sedation for CT imaging studies. Paediatr Anaesth. 2008 May;18(5):393-402. doi: 10.1111/j.1460-9592.2008.02451.x. Epub 2008 Mar 18. PMID 18363628
- [Background] Koroglu A, Teksan H, Sagir O, Yucel A, Toprak HI, Ersoy OM. A comparison of the sedative, hemodynamic, and respiratory effects of dexmedetomidine and propofol in children undergoing magnetic resonance imaging. Anesth Analg. 2006 Jul;103(1):63-7, table of contents. doi: 10.1213/01.ANE.0000219592.82598.AA. PMID 16790627
- [Background] Usher AG, Kearney RA, Tsui BC. Propofol total intravenous anesthesia for MRI in children. Paediatr Anaesth. 2005 Jan;15(1):23-8. doi: 10.1111/j.1460-9592.2004.01390.x. PMID 15649159
- [Background] Frankville DD, Spear RM, Dyck JB. The dose of propofol required to prevent children from moving during magnetic resonance imaging. Anesthesiology. 1993 Nov;79(5):953-8. doi: 10.1097/00000542-199311000-00013. PMID 8239013
- [Background] Levati A, Colombo N, Arosio EM, Savoia G, Tommasino C, Scialfa G, Boselli L. Propofol anaesthesia in spontaneously breathing paediatric patients during magnetic resonance imaging. Acta Anaesthesiol Scand. 1996 May;40(5):561-5. doi: 10.1111/j.1399-6576.1996.tb04488.x. PMID 8792885
- [Background] Evans RG, Crawford MW, Noseworthy MD, Yoo SJ. Effect of increasing depth of propofol anesthesia on upper airway configuration in children. Anesthesiology. 2003 Sep;99(3):596-602. doi: 10.1097/00000542-200309000-00014. PMID 12960543
- [Background] Litman RS, Weissend EE, Shrier DA, Ward DS. Morphologic changes in the upper airway of children during awakening from propofol administration. Anesthesiology. 2002 Mar;96(3):607-11. doi: 10.1097/00000542-200203000-00016. PMID 11873035
- [Background] Mathru M, Esch O, Lang J, Herbert ME, Chaljub G, Goodacre B, vanSonnenberg E. Magnetic resonance imaging of the upper airway. Effects of propofol anesthesia and nasal continuous positive airway pressure in humans. Anesthesiology. 1996 Feb;84(2):273-9. doi: 10.1097/00000542-199602000-00004. PMID 8602656
- [Background] Thompson JR, Schneider S, Ashwal S, Holden BS, Hinshaw DB Jr, Hasso AN. The choice of sedation for computed tomography in children: a prospective evaluation. Radiology. 1982 May;143(2):475-9. doi: 10.1148/radiology.143.2.7071350.
- [Background] Napoli KL, Ingall CG, Martin GR. Safety and efficacy of chloral hydrate sedation in children undergoing echocardiography. J Pediatr. 1996 Aug;129(2):287-91. doi: 10.1016/s0022-3476(96)70256-1. PMID 8765629
- [Background] Greenberg SB, Faerber EN, Aspinall CL, Adams RC. High-dose chloral hydrate sedation for children undergoing MR imaging: safety and efficacy in relation to age. AJR Am J Roentgenol. 1993 Sep;161(3):639-41. doi: 10.2214/ajr.161.3.8352124.
- [Background] Ronchera-Oms CL, Casillas C, Marti-Bonmati L, Poyatos C, Tomas J, Sobejano A, Jimenez NV. Oral chloral hydrate provides effective and safe sedation in paediatric magnetic resonance imaging. J Clin Pharm Ther. 1994 Aug;19(4):239-43. doi: 10.1111/j.1365-2710.1994.tb00680.x. PMID 7989402
- [Background] Hall JE, Uhrich TD, Barney JA, Arain SR, Ebert TJ. Sedative, amnestic, and analgesic properties of small-dose dexmedetomidine infusions. Anesth Analg. 2000 Mar;90(3):699-705. doi: 10.1097/00000539-200003000-00035. PMID 10702460

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propofol | Dexmedetomidine
Started | 30 | 30
Completed | 30 | 28 (Two of the original DEX group subjects were removed, due to receiving dexmedetomidine and propofol.)
Not Completed | 0 | 2
Not completed — Patients failed to reach sedation level | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Dexmedetomidine | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 8.8 [5.8 to 14.3] | 8.3 [4.7 to 16.1] | 8.6 [5.3 to 15.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 22 | 22 | 44
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Cross Sectional Area of the Pharyngeal Airway
Description: The primary outcome measures will be the cross sectional area of the pharyngeal airway of the patients measured at two levels soft palate (nasopharyngeal) and base of the tongue (retroglossal). Magnetic resonance images of the airway were obtained during low (1 mcg/kg/hr) and high (3 mcg/kg/hr) doses of DEX or low (100 mcg/kg/m) and high (200 mcg/kg/m) doses of Propofol. All were administered through an intravenous (IV) catheter.
Time Frame: during MRI within first 10 minutes of scanning
Measure: Median (95% Confidence Interval); unit: mm^2
Groups:
- Propofol: * Once an IV is in place, atropine 10 mcg/kg will be given. Loading dose of propofol 2 mg/kg will be administered over 2 minutes followed by a continuous infusion of propofol at rate of 100 mcg/kg/minute using a syringe pump (Low dose). Baseline airway images are obtained during this time.
  * If a subject moves during baseline images a bolus of Propofol 0.5 mcg/kg will be given over 10 seconds and infusion rate will be increased to 120 mcg/kg/hr. If the subject moves a second time the research study will be terminated and patient will be under care of clinical team.
  * After the initial set of airway images are obtained, a bolus dose of propofol 2 mcg/kg will be given over 2 minutes followed by an increase in the infusion rate to 200 mcg/kg/hr (high dose).
- Dexmedetomidine: * Once an IV is in place, atropine 10 mcg/kg will be given. Loading dose of dexmedetomidine 1 mcg/kg will be administered over 10 minutes followed by a continuous infusion of dexmedetomidine at rate of 1 mcg/kg/h using a syringe pump (low dose). Baseline airway images are obtained during this time.
  * If a subject moves during baseline images a bolus of DEX 0.5 mcg/kg will be given over 3 minutes and infusion rate will be increased to 1.5 mcg/kg/hr. If the subject moves a second time the research study will be terminated and patient will be under care of clinical team.
  * After the initial set of airway images are obtained, a 2 mcg/kg bolus of DEX will be given over 10 minutes followed by an increase in the infusion rate to 3 mcg/kg/hr (high dose).
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 30 | 28
mm^2
  Low Dose Sedative, Nasopharyngeal measurement | 239.9 [185.4 to 267.2] | 178.5 [148.5 to 222.4]
  High Dose Sedative, Nasopharyngeal measurement | 201.6 [148.9 to 291.7] | 235.4 [145.0 to 258.8]
  Low Dose Sedative, Retroglossal measurement | 115.1 [67.8 to 167.0] | 120.9 [63.6 to 179.5]
  High dose sedative, Retroglossal measurement | 108.1 [53.6 to 134.4] | 120.5 [50.1 to 178.4]

2. Secondary Outcome: Obstructive Index Until Recovery Room Discharge
Description: The Obstructive Index is a count of the obstructive apnea events per hour of sleep
Time Frame: During MRI and until recovery room discharge - approximately 30-250 minutes
Measure: Mean (Inter-Quartile Range); unit: Apnea events/hour of sleep
Groups:
- Mild OSA and Dexmedetomidine; Moderate OSA and Dexmedetomidine; Severe OSA and Dexmedetomidine: Patients were stratified by OSA severity as documented on the patient's sleep study report: mild, moderate, or severe. (Mild=obstructive index 1-5, Moderate= obstructive index >5-10, Severe=obstructive index>10)
  Additionally this patient was assigned to receive DEX.
- Mild OSA and Propofol; Moderate OSA and Propofol; Severe OSA and Propofol: Patients were stratified by OSA severity as documented on the patient's sleep study report: mild, moderate, or severe. (Mild=obstructive index 1-5, Moderate= obstructive index >5-10, Severe=obstructive index>10)
  Additionally this patient was assigned to receive Propofol.
Arm/Group | Mild OSA and Dexmedetomidine | Mild OSA and Propofol | Moderate OSA and Dexmedetomidine | Moderate OSA and Propofol | Severe OSA and Dexmedetomidine | Severe OSA and Propofol
Number analyzed (Participants) | 2 | 7 | 13 | 10 | 11 | 13
Apnea events/hour of sleep | 4.2 [3.4 to 4.9] | 3.0 [2.3 to 3.5] | 8.0 [7.4 to 8.6] | 8.0 [5.9 to 8.9] | 16.7 [14.1 to 23.3] | 17.1 [14.6 to 37.0]

3. Secondary Outcome: Respiratory Disturbance Index
Description: The respiratory disturbance index is a count of respiratory disturbance events per hour of sleep.
Time Frame: During MRI and until recovery room discharge - approximately 30-250 minutes
Measure: Mean (Inter-Quartile Range); unit: respir.disturbance events/hr of sleep
Arm/Group | Mild OSA and Dexmedetomidine | Mild OSA and Propofol | Moderate OSA and Dexmedetomidine | Moderate OSA and Propofol | Severe OSA and Dexmedetomidine | Severe OSA and Propofol
Number analyzed (Participants) | 2 | 7 | 13 | 10 | 11 | 13
respir.disturbance events/hr of sleep | 5.1 [4.8 to 5.4] | 3.2 [2.4 to 4.1] | 8.8 [7.7 to 9.8] | 7.1 [5.9 to 9.1] | 16.6 [14.3 to 19.6] | 25.2 [14.7 to 41.9]

4. Secondary Outcome: Needed Artificial Airway
Description: This is the count of the number of patients who needed an artificial airway.
Time Frame: During MRI and until recovery room discharge - approximately 30-250 minutes
Measure: Number; unit: Number of artifical airway events
Arm/Group | Mild OSA and Dexmedetomidine | Mild OSA and Propofol | Moderate OSA and Dexmedetomidine | Moderate OSA and Propofol | Severe OSA and Dexmedetomidine | Severe OSA and Propofol
Number analyzed (Participants) | 2 | 7 | 13 | 10 | 11 | 13
Number of artifical airway events | 0 | 1 | 1 | 1 | 2 | 5

5. Secondary Outcome: Room Air SpO2
Description: The patient's oxygen saturation on room air.
Time Frame: During MRI and until recovery room discharge - approximately 30-250 minutes
Measure: Mean (Inter-Quartile Range); unit: percentage of SpO2
Arm/Group | Mild OSA and Dexmedetomidine | Mild OSA and Propofol | Moderate OSA and Dexmedetomidine | Moderate OSA and Propofol | Severe OSA and Dexmedetomidine | Severe OSA and Propofol
Number analyzed (Participants) | 2 | 7 | 13 | 10 | 11 | 13
percentage of SpO2 | 87.2 [86.7 to 87.7] | 88.0 [83.0 to 91.0] | 86.3 [84.8 to 87.5] | 89.0 [87.0 to 93.0] | 84.0 [77.0 to 88.8] | 88.0 [80.4 to 88.2]

ADVERSE EVENTS:
Arm/Group | Propofol | Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Failure to standardize mouth opening, due to stimulation of the subject during manipulation of the mouth No baseline measurements were obtained while awake Many patients had Downs syndrome so the results may not apply across all patients with OSA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes